CLINICAL TRIAL: NCT00780442
Title: D-Cycloserine and Cue Exposure in Cocaine-Dependent Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Professor of Psychiatry and Behavioral Sciences, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HR#16454
Record Dates: First submitted 2008-10-23; First posted 2008-10-27 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Cocaine Use Disorders
Keywords: substance related disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DCS (Experimental): D-Cycloserine 50 mg is a partial glutamate agonist. Participants received DCS prior to cocaine cue exposure sessions.
  Interventions: Drug: D-cycloserine
- Placebo (Placebo Comparator): Saline comparator. Participants received placebo prior to cocaine cue exposure sessions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — 50 mg DCS
  Arms: DCS
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
In summary, this pilot study will explore the use of an innovative pharmacologic approach to the treatment of substance dependence through the facilitation of extinction of response to cocaine-conditioned cues in cocaine-dependent individuals. If DCS proves successful in this preliminary study, a controlled treatment trial will be planned. This novel approach could have implications for the treatment of multiple substance use disorders including methamphetamine, marijuana and opiate dependence.

DETAILED DESCRIPTION:
Cocaine dependence remains a serious problem in the US today and in spite of two decades of intense research, efficacious pharmacotherapeutic treatments have not been identified. Cocaine-associated environmental cues can elicit drug craving and exposure to cocaine-related cues is likely to be involved in relapse. Emerging data supports the role of glutamate in extinction of associative learning in animal models of rear-conditioning and clinical studies of exposure treatment for anxiety disorders. A recent study demonstrated DCS acceleration of cocaine-induced conditioned place preference in rats. Exploration of DCS in facilitating extinction of response to drug-related cues in humans is needed. The proposed study will extend these innovative and promising findings from the basic science arena and anxiety disorders field in a proof of concept investigation of DCS facilitation of extinction of response to cocaine-related cues in a human laboratory paradigm.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Subjects must meet DSM-IV criteria for current cocaine dependence. Subjects may meet criteria for abuse, but not dependence on any other substance within the past 60 days with the exception of nicotine. Because of the high comorbidity of cocaine and nicotine dependence, excluding nicotine dependence would seriously compromise the feasibility of recruitment. Nicotine use immediately prior to the testing session will be controlled. Alcohol has also been known to affect HPA function, however to enhance recruitment efforts individuals with alcohol dependence or abuse will be included in the study if they do not require medically supervised detoxification.
3. Use of one of the following methods of birth control by female subjects: barrier methods (diaphragm or condoms with spermicide or both), surgical sterilization, use of an intra-uterine contraceptive device, or complete abstinence from sexual intercourse.
4. Subjects must live within a 50-mile radius of our research program and have reliable transportation.
5. Subjects must consent to remain abstinent from all drugs of abuse (except nicotine or alcohol) for 24 hours immediately prior to the GCRC admission.
6. Subjects must consent to random assignment to the DCS vs. placebo conditions.

Exclusion Criteria:

1. Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
2. Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect heart rate or skin conductance measurement.
3. Individuals with creatinine clearance of 1.2 or greater as DCS is renally excreted.
4. Subjects with a history of or current psychotic disorder, current major depressive disorder, bipolar affective disorder or a severe anxiety disorder as these may impact cue reactivity.
5. Subjects who are unwilling or unable to maintain abstinent from alcohol and other drugs of abuse (except nicotine) for 24 hours days prior to the cue procedure.
6. Subjects meeting DSM-IV criteria for substance dependence (other than nicotine or cocaine as appropriate) within the past 60 days.
7. Subjects currently taking B-blockers, anti-arrythmic agents, psychostimulants or any other agents known to interfere with heart rate and skin conductance monitoring.
8. Known or suspected hypersensitivity to DCS.
9. Individuals taking medications that could adversely interact with study medications, including, but not limited to ethionamide, isoniazid, or amino acid supplements.
10. Subjects with a history of epilepsy or seizure disorder.
11. Subjects with significant liver impairment as DCS may increase serum transaminases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee L McRae, Pharm.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- D-cycloserine: Participants received DCS prior to cocaine cue exposure sessions.
- Placebo: Participants received placebo prior to cocaine cue exposure sessions.
Period: Overall Study
Arm/Group | D-cycloserine | Placebo
Started | 12 | 15
Completed | 12 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine | Placebo | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 15 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Craving Scale
Description: Scale assess cocaine craving following cocaine cue exposure after two administrations of DCS. Subjects rate craving on a scale from 0-10 with 0 indicating "Not at all" and 10 indicating "Extremely".
Time Frame: Immediately following cue exposure
Population: Cocaine dependent individuals
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 12 | 15
Units on a scale | 4.33 (3.98) | 3.13 (2.92)

ADVERSE EVENTS:
Arm/Group | D-cycloserine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes